CLINICAL TRIAL: NCT01568606
Title: Safety of Body Composition Analysis Using Bioimpedance in Heart Failure Patients With Implantable Cardioverter Defibrillators (ICDs)
Brief Title: Safety of Body Composition Analysis in Heart Failure Patients With Implantable Cardioverter Defibrillators (ICDs)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Tamara Horwich, Dr. Tamara Horwich, M.D., M.S., University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: UCLA M-IRB1 # 10-001055
Record Dates: First submitted 2011-08-15; First posted 2012-04-02 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure; Obesity
Keywords: Heart Failure; Obesity; Implantable Cardioverter Defibrillator
MeSH Terms: conditions — Heart Failure; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Body Composition Analysis InBody Scale (Experimental)
  Interventions: Device: Body Composition Analysis InBody Scale

INTERVENTIONS:
Device: Body Composition Analysis InBody Scale — Patients will have their ICD interrogated using a pacemaker Programmer specifically designed from one of the 4 pacemaker manufacturers: St. Jude, Medtronic, Guidant, and Biotronik. Depending on the type of pacemaker, interrogation can be done either wirelessly or by placing a wand over the pacemaker. The ICD will be turned to a "monitor-only" mode to disable risk of ICD shock by the supervising electrophysiologist. Patient will be asked to step on the InBody 520 scale to have their body composition analyzed. Patient will continue to have their ICD actively monitored. Analysis will take approximately 30 - 50 seconds. At the end of analysis, ICD device will be returned to default settings by supervising electrophysiologist.
  Other Names: Body Composition Analysis InBody 520 Scale

SUMMARY:
The purpose of this study is to define the safety of using bioimpedance for analysis of body composition in heart failure patients with ICD devices. The Biospace America InBody 520 scale, using direct segmental multifrequency bioimpedance, will be utilized to assess patients' fat mass, lean muscle mass, and edema status.

Although the Biospace America InBody 520 scale is routinely used to analyze body composition in various settings including the Ahmanson-UCLA Cardiomyopathy clinic, due to theoretical concerns of safety, bioimpedance has not been routinely used in patients with ICDs. The investigators hope that this study will allow us to routinely analyze body composition in heart failure patients with ICDs, information which can be used to help guide dietary, exercise, and medical prescriptions for the investigators heart failure patients.

DETAILED DESCRIPTION:
Up to one half of heart failure (HF) patients are overweight and obese, as measured by body mass index (BMI). Comprehensive body composition assessment utilizing bioimpedance scales wuch as Biospace America InBody 520 scale, can give accurate measurements of fat mass, lean muscle mass, and edematous water weight. Body composition analysis is routinely used in many clinical settings, including the Ahmanson-UCLA Cardiomyopathy Center. However, bioimpedance scales are generally not used in patients with implantable cardioverter-defibrillators (ICDs), a group that represents a majority of our HF patient population. The safety of InBody 520 technology - direct segmental multifrequency (5, 100, 500 KHz) bioimpedance analysis - in patients with ICDs has not been formally evaluated. There is a theoretic concern that the ICD may misinterpret the applied currents for a cardiac arrhythmia and possibly cause a discharge from the ICD. However, there has been no documentation of any adverse events in patients with ICDs using the InBody 520 or other bioimpedance scales. Furthermore, thoracic bioimpedance analysis (BioZ ICG, 70 Khz) has been documented to be successfully utilized without adverse effects in patients with HF and ICDs. This study will define the safety of using the InBody 520 scale for analysis of body composition in patients with ICD devices. Subjects with HF and and ICD will have their ICD interrogated and continually monitored by an electrophysiologist before, during, and after the 30-50 seconds of bioimpedance analysis, which involves standing on the InBody 520 scale. If there is any suggestion of the ICD interpreting applied frequencies as a cardiac arrhythmia, the patient will be removed from the scale and the electrophysiologist will simultaneously temporarily deactivate their ICD device to prevent discharge. Twenty subjects (from the following four ICD companies: Medtronic, St. Jude, Guidant, and Biotronik) will participate in our study.

ELIGIBILITY:
Inclusion Criteria:

* HF patients of any etiology who currently have an implanted ICD

Exclusion Criteria:

* patients who are non-ambulatory
* have a physical disability making them unable to stand on the InBody
* those who are above the height and weight maximums for the device [Height > 220cm (7'2.6''), Weight > 250kg (551lb)]
* those who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Horwich, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- Ahmanson-UCLA Cardiomyopathy Center, Los Angeles, California, United States

REFERENCES:
- [Result] Buch E, Bradfield J, Larson T, Horwich T. Effect of bioimpedance body composition analysis on function of implanted cardiac devices. Pacing Clin Electrophysiol. 2012 Jun;35(6):681-4. doi: 10.1111/j.1540-8159.2012.03377.x. Epub 2012 Mar 27. PMID 22452409

RESULTS

PARTICIPANT FLOW:
Groups:
- Body Composition Analysis InBody Scale: Subjects with HF and ICD had their ICD interrogated and continually monitored by an electrophysiologist before, during, and after the 30-50 seconds of bioimpedance analysis, which involves standing on the InBody 520 scale. Outcome measure was assessed during a one day visit. There is no further follow-up.
Period: Overall Study
Arm/Group | Body Composition Analysis InBody Scale
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Body Composition Analysis InBody Scale
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Arrhythmia as Detected by ICD
Description: Subjects with HF and ICD had their ICD interrogated and continually monitored by an electrophysiologist before, during, and after 30-50 seconds of bioimpedance analysis, which involves standing on the InBody 520 scale. Outcome measure was assessed during a one day visit. There is no further follow-up.
Time Frame: 1 day, on day of study ICD interrogated and continually monitored before, during, and after 30-50 seconds of bioimpedance analysis
Measure: Number; unit: participants
Groups:
- Body Composition Analysis InBody Scale: Subjects with HF and ICD had their ICD interrogated and continually monitored by an electrophysiologist before, during, and after the 30-50 seconds of bioimpedance analysis, which involves standing on the InBody 520 scale.
Arm/Group | Body Composition Analysis InBody Scale
Number analyzed (Participants) | 20
participants | 0

ADVERSE EVENTS:
Time Frame: 1 day, on day of study ICD interrogated and continually monitored before, during, and after 30-50 seconds of bioimpedance analysis
Arm/Group | Body Composition Analysis InBody Scale
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

LIMITATIONS AND CAVEATS:
Due to small sample, we cannot exclude rare BIA-ICD interactions. Results may not be generalizable to other devices or BIA systems that utilize different frequencies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes